CLINICAL TRIAL: NCT02634892
Title: Pressure Redistributing Overlay With Targeted Cooling Technology (PRO-TECT) for Pressure Ulcer Prevention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: David Brienza (Other)
Responsible Party: Sponsor-Investigator, David Brienza, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO14120116
Record Dates: First submitted 2015-12-06; First posted 2015-12-18 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Pressure Ulcer
Keywords: Sacral; Overlay Mattress; Cooling
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care (SOC) (No Intervention): Patients receive usual or standard of care regarding management of early stage pressure ulcers
- SOC plus PRO-TECT (Experimental): Patients receive usual or standard of care plus the addition of PRO-TECT.
  Interventions: Device: PRO-TECT

INTERVENTIONS:
Device: PRO-TECT — Patient will be placed on ROHO SOFFLEX2 mattress with has been modified with gel cushions in the sacral region for heal dissipation by standard closed system cooling pad
  Arms: SOC plus PRO-TECT

SUMMARY:
Objective - To demonstrate the efficacy of the pressure redistributing cooling mattress overlay compared to usual care in mitigating the progression of early pressure ulcers in critically ill (ICU) patients via a prospective randomized human clinical trial.

Specific Aim - The clinical trial will evaluate the efficacy and safety of the PRO-TECT ™ mattress overlay in ICU patients who have already developed early pressure ulcers (Stage 1 and 2) and preventing further progression to more severe pressure ulcers (Stage 3 and 4) as well as potential faster regression (i.e. healing of Stage 1 and 2 pressures).

DETAILED DESCRIPTION:
To demonstrate the efficacy of the pressure redistributing cooling mattress overlay for prevention of pressure ulcers in critical care units, a prospective randomized human clinical trial will be performed. The trial will use functionally equivalent test overlays. The initial pilot clinical trial will evaluate the efficacy and safety of the PRO-TECT ™ mattress overlay in ICU patients who have already developed early pressure ulcers (Stage 1 and 2) and preventing further progression.

The trial will be performed in UPMC ICUs by enrolling patients age 18 or older with Stage 1 and Stage 2 sacral/coccyx pressure ulcers. The trial will consist of 2 arms: 1) current usual care (UC) vs. 2) UC + targeted cooling overlay mattress (TCOM). Exclusion criteria will include anticipated ICU length of stay < 3 days, patients initially designated for specialty overlay/bed for pulmonary or bariatric diagnoses, patients with a Stage 3 or 4 or unstageable pressure ulcer on the sacrum.

The UC group will receive current UPMC ICU guideline-based care with daily assessments for sacral pressure ulcers. Nursing care guidelines will be applied including frequent patient turning, pressure alleviation, moisture control, and friction relief applications. Patients in this group may receive a specialty bed or overlay mattress without cooling if recommended by wound care specialist. The TCOM group will receive UC plus overlay mattress with targeted sacral cooling.

Wound care as well as assessment will be performed daily by the non-wound care nurses ( ie. ICU nurse while under ICU care and Floor nurses while under non-ICU care) as part of their regular daily assessment for both non-target cooling and targeted cooling patients. Wound care specialist will assess the wound on Mon/Wed/Fri for any progression or deterioration of the wounds. These wound care nurses are specialty trained in stage decubitus as well as recommending changes in care to promote healing. Additionally they will record the data as part of their routine care of patient with wounds. Theses types of wound assessments are best performed every 2-3 days in order to see any significant change of therapy and data will be recorded.

Data collected on Monday, Wednesday and Friday of each week including Braden score, pressure ulcer stage, healing progression (or deterioration) with measurements (e.g., size), and evidence of infection. Additionally, frequency of patient reposition will be recorded and if not, documentation of justification will be provided. Other data collected will include demographics, vitals, comorbidities, length of times (prior incapacitation at home or nursing facility, transport, emergency department, operative room), ventilation and oxygenation requirement, ventilator days, ICU LOS, need for dialysis, vasopressors, and labs including nutritional labs. Data will be collected until study endpoint of discharge from hospital. Final cost analysis will be performed to compile a cost-benefit of each arm. Accrual will be 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-100 years of age
* Patients with Stage 1 or 2 pressure ulcers

Exclusion Criteria:

* Patients < 18 years old
* Patients admitted directly to non-critical care beds
* Patients with undetermined stage or late stage (3 or 4) pressure ulcers
* Patients with Raynauds disease
* Patients with spina bifida

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Final Pressure Ulcer Stage | at each patient discharged from acute care hospital setting, usually 2-4 weeks
  Measure of the severity of the pressure ulcer at the time of discharge

CONTACTS AND LOCATIONS:
Overall Officials: David M Brienza, PhD, Principal Investigator — University of Pittsburgh